CLINICAL TRIAL: NCT03737201
Title: Ozone Application in Stepwise Excavation
Brief Title: Influence of Ozone Application in Stepwise Excavation Procedure of Primary Molars With Deep Carious Lesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Merve AKCAY, Assoc. Prof., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 213S004-2
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Deep Caries; Ozone
Keywords: ozone; Deep Carious Lesion; Primary Molars
MeSH Terms: interventions — Ozone; chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: randomized, three-arm parallel, two-blinded clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ozone (Experimental): Thirty five molar teeth with deep caries lesion were selected to apply two-visit indirect pulp therapy with ozone. The peripheral demineralized dentin and the superficial necrotic dentin were completely removed, and left some caries at the central part. The cavity was exposed to gaseous ozone for 60 seconds, with an ozone delivery system. The remaining caries dentin was covered with calcium hydroxide base material and cavity sealed with glass ionomer cement to reopen 4 months later.
  Interventions: Other: ozone
- chlorhexidine digluconate (Active Comparator): Thirty five molar teeth with deep caries lesion were selected to apply two-visit indirect pulp therapy with chlorhexidine digluconate. The peripheral demineralized dentin and the superficial necrotic dentin were completely removed, and left some caries at the central part. Following the excavation, 2% chlorhexidine digluconate was applied to the cavity for 60 seconds using a brush. According to the manufacturer instructions, puddled solution was removed with a new brush without dry to leave site moist. The remaining caries dentin was covered with calcium hydroxide base material and cavity sealed with glass ionomer cement.
  Interventions: Other: chlorhexidine digluconate
- control (Active Comparator): Thirty five molar teeth with deep caries lesion were selected to apply conventional two-visit indirect pulp therapy (control). The peripheral demineralized dentin and the superficial necrotic dentin were completely removed, and left some caries at the central part. The remaining caries dentin was covered with calcium hydroxide base material and cavity sealed with glass ionomer cement.
  Interventions: Other: Control

INTERVENTIONS:
Other: ozone — In the two-visit indirect pulp therapy, due to reduce the number of bacteria remaining in the cavity, the antimicrobial agents can be used as cavity disinfectants such as ozone.
  Arms: ozone
Other: chlorhexidine digluconate — In the two-visit indirect pulp therapy, due to reduce the number of bacteria remaining in the cavity, the antimicrobial agents can be used as cavity disinfectants such as chlorhexidine digluconate.
  Arms: chlorhexidine digluconate
Other: Control — without any cavity disinfectant
  Arms: control

SUMMARY:
Purpose: The purpose of this study was to investigate the clinical and microbiological effectiveness of the ozone application in stepwise excavation of primary molars.

Methods: This study was conducted in vivo conditions with 105 lower primary second molars that had deep caries lesions with the risk of pulpal exposure. The teeth were randomly divided into three groups: Conventional stepwise excavation without any disinfectant, 2% chlorhexidine digluconate(CHX) and ozone application. In four different stages (after; initial excavation, ozone/CHX application, four months, final excavation), dentine samples were collected for microbiological analysis of mutans streptococci, lactobacilli and total number of colony forming units. Clinical changes as dentine colour, humidity, consistency were recorded. The data were analysed by Mann-Whitney U, Friedman and chi-square test.

DETAILED DESCRIPTION:
Informed consent including possible risks, discomforts and benefits about the procedure were obtained from all parents of the young patients.

The required sample size for this study was 35 in each subgroup (82 percent power, two-sided five percent significance level) for the detection of a significant difference. This study was conducted on 105 patients aged 6 to 10 years (59 girls, 46 boys) who attended the Pediatric Dentistry Department. None of the patients included in the study were medically compromised. Each patient had one mandibular second primary molar with deep carious lesion and pulp perforation risk. All teeth with deep carious lesions were examined clinically and radiographically.

The following inclusion criteria were used;

* Active carious lesion in deep dentine of primary second molars,
* Absence of clinical symptoms of irreversible pulpitis such as spontaneous pain or longtime pain against thermal and chemical stimuli,
* Absence of sensitivity to percussion or palpation, pathological mobility, swelling or fistula any discoloration except for carious lesion.
* Absence of any interradicular lesions, periapical radiolucency, pathological resorptions and pulpal calcifications.

A randomized, controlled, clinical trial was designed in a sample of 105 primary molars (35 teeth in each group) as three treatment groups: Step-wise excavation without any disinfectant (control group), step-wise excavation with CHX application (positive control group), and step-wise excavation with gaseous ozone application (experimental group).

All procedures were performed by one investigator. After mandibular anesthesia of the tooth, rubber dam isolation was provided. Carious enamel, lateral walls of the cavity and necrotic dentin was removed with carbide burs. Removal of carious dentin was performed with dentin excavators and low speed-burs, and left some caries at the central part. It was decided to leave potentially mineralizable affected dentin by hand sensitivity. Following the same procedures, the teeth were randomly divided into 3 groups (n=35):

Control Group: After partial removal of carious dentin, calcium hydroxide [Ca(OH)2] base material (Dycal; Dentsply International Milford, USA) was placed on the remaining carious dentin without applying any cavity disinfectants.

Positive Control Group: After partial removal of carious dentin, 2% CHX solution (Cavity Cleanser, Bisco, USA) was applied to the cavity for 60 s with an applicator brush for disinfection procedure. According to the manufacturer instructions, puddled solution was removed with a new brush without dry to leave site moist. Then, Ca(OH)2 base (Dycal; Dentsply) was placed on the remaining carious dentin.

Experimental Group: After partial removal of carious dentin, ozone gas (Heal ozone, KaVo Dental, Germany) with the concentration of 2100 ppm was applied to the cavity for 60 s for disinfection procedure. Ozone production stopped if the airtight seal over the tooth was broken during treatment, therefore, silicon caps were selected according to the size of each tooth. And Ca(OH)2 base was placed on the remaining carious dentin.

All the teeth were then temporarily sealed with glass ionomer cement and coating agent. After 4 months, radiographic and clinical examinations were repeated. Following rubber dam isolation and anesthesia, temporary fillings were removed. Removing of Ca(OH)2 on the remaining carious dentin was carefully performed with excavators. Subsequent to this procedure, remaining demineralized dentin was completely removed in all groups. Floor of the cavity was then covered with Ca(OH)2 base material (Dycal; Dentsply/Caulk) and glass ionomer lining. The cavities were then restored with composite resin after the 2-stages self-etch bond application.

Microbiological analysis:

During these procedures dentin samples were collected with a sterile carbide bur #14 from each group for microbiological analyses.

Clinical photograph was taken with dental explorers pointing to ensure that all samples were collected from the same site in all following stages. The dentine samples were collected enough to fill the slots of a sterile No.14 round carbide bur and the respective samples were placed into 1 ml thiogluconate medium then transported to the microbiology laboratory in 2 hours to be analyzed for the mutans streptococci, lactobacilli and the total number of colony forming units (CFU).

The samples were homogenized on a vortex mixer for 15 seconds under laboratory conditions. Mitis Salivarius agar as the selective medium for Streptococcus mutans, rogosa agar for Lactobacilli and Brain Hearth agar supplemented 5% blood for the total number of CFU were used. Tenfold dilution were plated onto agars and incubated anaerobically for 48 hours and the colonies were counted on the convenient dilution.

Clinical Evaluation For the clinical analysis, the colour, consistency and humidity of the dentine were also recorded during taking microbiological samples.

Color findings classifications were recorded according to following criteria: Light yellow, yellow, light brown, dark brown, black. Classification of dentin consistency was determined by probing and criteria were "very soft", " "soft", "moderate hard" and "hard". Dentin humidity was recorded as "wet" and "dry". Accordingly, the dentine was probed and if moisture leakage occurred, it was classified as wet or if it did not then it would be classified as dry.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, vital and asymptomatic lower primary molars with deep caries lesions considered likely to result in pulp exposure if they were treated by a single and terminal excavation
* Positive pulp sensibility tested by an electric pulp tester and cold stimulation,
* Mild discomfort from chemical and thermal stimuli,
* Cooperative children and parents willing to follow the instructions and report for follow-up.

Exclusion Criteria:

* Signs of irreversible pulpitis (spontaneous pain, prolonged pain response etc.)
* The presence of percussion or palpation sensitivity, pathological mobility, or infection symptoms like fistula or abscess or discoloration in the clinical examination,
* Absence of normal lamina dura and periodontal range, presence of lesion, internal or external resorption or calcification in or around the root in the radiological examination,
* Children with special health care needs.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Changes microbiological count: from baseline to 4 months | Baseline and Four months later
  Mutans streptococci counts were calculated.
Changes microbiological count: from baseline to 4 months | Baseline and Four months later
  Lactobacilli counts were calculated.
Changes microbiological count: from baseline to 4 months | Baseline and Four months later
  Total number of colony forming units counts were calculated.

SECONDARY OUTCOMES:
Changes characteristics of the dentin humidity: from baseline to 4 months | Baseline and Four months later
  Dentine was probed and if moisture leakage was occurred, it was classified as wet or if did not it would be classified as dry.
Changes characteristics of the dentin consistency: from baseline to 4 months | Baseline and Four months later
  The consistency of dentin was determined by probing and classified as; very soft, soft, medium hard and hard.
Changes characteristics of the dentin color: from baseline to 4 months | Baseline and Four months later
  The colour of dentin was classified as, light yellow, yellow, light brown, dark brown/black.

IPD SHARING:
Plan to Share IPD: No